CLINICAL TRIAL: NCT05860439
Title: Long-term Follow-up of Sclerotherapy of Reticular Veins and Telangiectasias
Brief Title: Lower Limb Sclerotherapy of Reticular Veins and Telangiectasias
Status: Completed | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Other Study IDs: UPECLIN233283
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Telangiectasis
Keywords: Sclerotherapy; Veins; Telangiectasias; Hyperpigmentation
MeSH Terms: conditions — Telangiectasis; Hyperpigmentation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Telangiectasias Group - Polidocanol 0,2% + Hypertonic Glucose 70% (PDHG): Previously treated with PDHG, no new interventions were performed.
  Interventions: Procedure: Polidocanol 0,2% + Hypertonic Glucose 70% (PDHG)
- Telangiectasias Group - Hypertonic Glucose 75% (HG): Previously treated with HG, no new interventions were performed.
- Reticular Veins Group (PG3T) - Polidocanol 0,2% + Hypertonic Glucose 70% (PDHG): Previously treated with PDHG, no new interventions were performed.
  Interventions: Procedure: Polidocanol 0,2% + Hypertonic Glucose 70% (PDHG)
- Reticular Veins Group (PG3T) - Hypertonic Glucose 75% (HG): Previously treated with HG, no new interventions were performed.

INTERVENTIONS:
Procedure: Polidocanol 0,2% + Hypertonic Glucose 70% (PDHG) — Patients previously treated were reassessed for long-term follow-up.
  Other Names: Hypertonic Glucose 75% (HG)
  Groups: Reticular Veins Group (PG3T) - Polidocanol 0,2% + Hypertonic Glucose 70% (PDHG); Telangiectasias Group - Polidocanol 0,2% + Hypertonic Glucose 70% (PDHG)

SUMMARY:
A long-term follow-up cohort study of patients that were assigned in two previous studies to compare the clinical results of sclerotherapy of telangiectasias and reticular veins of lower limbs using 0.2% polidocanol diluted in 70% hypertonic glucose (PDHG) vs 75% hypertonic glucose (HG) alone.

All women, previously treated as aforementioned, were invited to be reevaluated regarding late maintenance and pigmentation over two years of follow-up.

No new treatments were applied to the cohort.

ELIGIBILITY:
Inclusion Criteria:

* All patients that concluded the participation of 60 days in both primary studies were invited to reevaluate the actual status of treatment (maintenance of treated vessels) and late complications (pigmentation and matting).

Exclusion Criteria:

* Patients who did not agree to be reassessed;
* Patients who were not found after all available forms of contact had been tried;
* Patients who went through any kind of intervention on the area of interest in lower limbs between the end of the intervention and the reevaluation for long-term follow-up.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women between 18 and 90 years, with lower limb telangiectasias or reticular veins treated in previous studies with polidocanol plus hypertonic glucose or hypertonic glucose.
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Length of Telangiectasias in Centimeters | 730 days
  Total length of telangiectasias at day 730 for comparison with day 60 and assessment of disease relapse.

SECONDARY OUTCOMES:
Length of Hyperchromia in Centimeters | 730 days
  Total length of hyperchromic stains at day 730 for comparison with day 60 and assessment of reversion.
Length of Matting in Centimeters | 730 days
  Total length of matting neovascularization at day 730 for comparison with day 60 and assessment of reversion.

CONTACTS AND LOCATIONS:
Locations (1):
- Sao Paulo State University Botucatu Campus, Botucatu, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No